CLINICAL TRIAL: NCT07335705
Title: Analysis of Factors Influencing the Quality of Bowel Preparation Before Colonoscopy in IBD Patients: A National Multicenter Prospective Study
Brief Title: Analysis of Factors Influencing the Quality of Bowel Preparation Before Colonoscopy in IBD Patients
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, professor, Changhai Hospital
Other Study IDs: CHEC2025-448
Record Dates: First submitted 2025-12-08; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: IBD (Inflammatory Bowel Disease); Colonoscopy; Colonoscopy: Bowel Preparation
Keywords: IBD; Colonoscopy; Bowel preparation
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort for Bowel Preparation in IBD Patients: Patients aged 18 years or older diagnosed with Inflammatory Bowel Disease (IBD) and scheduled for a colonoscopy, who undergo standard bowel preparation procedures followed by colonoscopy examination and questionnaire completion.
  Interventions: Other: Standard Pre-colonoscopy Bowel Preparation Protocol

INTERVENTIONS:
Other: Standard Pre-colonoscopy Bowel Preparation Protocol — This involves standard clinical instructions including a low-residue diet prior to colonoscopy and the administration of bowel cleansing agents (e.g., Polyethylene Glycol) according to the split-dose regimen as per each participating center's routine practice. The timing, dosage, and specific agent used follow existing institutional guidelines.

SUMMARY:
The primary objectives of this project are twofold. On the one hand, it aims to investigate the current status of bowel preparation protocols and their quality in IBD patients undergoing colonoscopy, particularly focusing on the implementation of these protocols across hospitals following the release of the 2023 bowel preparation guidelines. This will further standardize and optimize bowel preparation practices in China. On the other hand, the project seeks to identify and examine various risk factors contributing to poor bowel preparation quality in IBD patients, analyze their correlation with bowel preparation scores, and develop a risk prediction model for failed bowel preparation. This will provide a theoretical foundation for formulating personalized bowel preparation regimens tailored to individual patient conditions in the future.

DETAILED DESCRIPTION:
Step 1: During the issuance of a colonoscopy order, outpatient/ward physicians conduct preliminary screening and introduction to potential participants. Alternatively, recruitment may take place during follow-up in the recovery room or ward after the patient completes the colonoscopy (must be within 7 days post-procedure to reduce recall bias). Provide detailed explanations of the study content, risks, and benefits to potential subjects.

Step 2: Ensure that the patient fully understands the study, and then proceed to sign the "Informed Consent Form."

Step 3: Patients complete the "Questionnaire on Factors Influencing Bowel Preparation in IBD Patients." The questionnaire covers two main aspects: First, potential risk factors that may affect the quality of bowel preparation, including BMI, history of abdominal surgery, history of diabetes, history of diarrhea or constipation, stool characteristics, etc. Second, the specific bowel preparation protocol, including pre-colonoscopy diet, type of bowel cleansing agent used, dosage, interval between completion of medication and start of colonoscopy (waiting time), timing of medication intake, etc. Finally, the researcher records the bowel preparation quality score and colonoscopy results, including Boston Bowel Preparation Scale scores for each intestinal segment, colonoscopic diagnosis, endoscopic disease activity scores, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, of any gender, scheduled for colonoscopy;
* Patients diagnosed with Inflammatory Bowel Disease (IBD) according to the 2023 edition of the Guidelines for the Diagnosis and Treatment of Inflammatory Bowel Disease;
* Voluntary participation in this study and provision of signed informed consent.

Exclusion Criteria:

* History of acute myocardial infarction (within the past 6 months), severe cardiac, hepatic, or renal insufficiency, or psychiatric disorders;
* Current use of anticoagulants (e.g., aspirin, warfarin) or presence of coagulation disorders;
* Pregnant or lactating women;
* Acute intestinal infection within the past 2 weeks;
* History of colorectal tumors, familial adenomatous polyposis, or Peutz-Jeghers syndrome;
* History of intestinal obstruction, perforation, stenosis, or any other condition preventing completion of the examination;
* Severe hearing impairment, cognitive dysfunction, or inability to cooperate with the survey;
* Individuals already enrolled in this study who schedule a repeat colonoscopy;
* Currently participating in another clinical observational trial or having participated in any other clinical trial within the past 60 days;
* Refusal to sign the written informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients (aged ≥18 years) diagnosed with Inflammatory Bowel Disease (IBD) according to the 2023 Chinese guidelines, who are scheduled to undergo a colonoscopy
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
adequate bowel preparation rate | The adequate bowel preparation rate can be assessed immediately upon completion of colonoscopy
  Proportion of subjects with Boston Bowel Preparation Scale (BBPS) scores ≥ 2 in all bowel segments.

SECONDARY OUTCOMES:
Patient Satisfaction | immediately upon completion of colonoscopy
  Patient satisfaction is rated on a 5-point Likert scale ranging from 0 (very dissatisfied) to 5 (very satisfied), with patients rating their satisfaction regarding the entire bowel preparation process from the day before to immediately before the colonoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China